CLINICAL TRIAL: NCT06857357
Title: Evaluation of Kinesiophobia in Patients With Headache Using the Tampa Kinesiophobia Scale Modified for Headache: Turkish Version, Validity and Reliability Study
Brief Title: Tampa Kinesiophobia Scale Modified for Headache
Acronym: Kinesiophobia
Status: Completed | Type: Observational
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Dilara Onan, Assistant Professor, Bozok University
Other Study IDs: 2024-GOKAEK2413_2024.11.20_190
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Migraine
Keywords: Migraine; kinesiophobia
MeSH Terms: conditions — Migraine Disorders; Kinesiophobia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — The Tampa Kinesiophobia Questionnaire is a 17-question questionnaire that assesses avoidance of injury and fear of movement. The scale is scored using a Likert scale (1 = Strongly disagree, 4 = Strongly agree). Items 4, 8, 12 and 16 are reversed to calculate the total score of the scale. The total score is between 17 and 68. As the score of the person increases, it is understood that their kinesiophobia is high. A total score higher than 37 is considered as high kinesiophobia. However, since not every item of the questionnaire addresses patients with headache in this study, some questions were removed, some questions were edited and some questions were added to create a kinesiophobia questionnaire for headache. The newly created questionnaire consists of 23 items. Again, it is scored using a Likert scale with "1 = Strongly disagree, 4 = Strongly agree". As the score increases, it is understood that the level of kinesiophobia is high.

SUMMARY:
Tampa Kinesiophobia Scale is a scale that has been validated and reliable in individuals with low back pain in the Turkish population and evaluates fear of movement due to the risk of triggering pain. Especially for migraine headache, patients have complaints about movement and fear of movement, and in addition, according to the International Classification of Headache Disorders, 3rd Edition criteria, the item of aggravation with physical activity is considered as a diagnostic criterion. Migraine patients may theoretically start their attacks due to hypocretin neuropeptide and lactate metabolism dysfunction. It has been stated that calcitonin gene-related peptide (CGRP), which is released during migraine attacks, is also released during exercise and intense physical activity and can trigger attacks. Therefore, patients avoid physical activity and exercise. It has been stated that movements that do not require effort can also trigger attacks in migraine patients. The aim of this study is to investigate the validity and reliability of the Tampa Kinesiophobia Scale for Headache in patients with migraine for the Turkish population. The potential relationships between the scale and the beliefs about headache intensity, disability, headache impact, anxiety and depression will also be evaluated and whether the characteristics of the three types of headaches are similar or different from kinesiophobia will be investigated.

Hypothesis:

H0: The Tampa Kinesiophobia Scale for Headache is not valid and reliable for the Turkish population in patients with migraine H1: The Tampa Kinesiophobia Scale for Headache is valid and reliable for the Turkish population in patients with migraine

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with episodic/chronic migraine,
* Being between the ages of 18-70,
* Being able to read, speak, understand and write Turkish in order to understand and correctly answer the items/questions of the surveys and scales.

Exclusion Criteria:

* Having a diagnosis of episodic/chronic migraine,
* Having a history of any systemic disease such as malignant, inflammatory, acute fracture, surgery, neurological, psychological, or rheumatological.
* Not being able to read Turkish.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-70 who applied to neurology departments of Mersin University, Gazi University, Zonguldak Bülent Ecevit University, Kütahya Health Sciences University, Gaziantep City Hospital, Silivri State Hospital, Trakya University, and Elite Research and Surgery Hospital and who were diagnosed with episodic/chronic migraine according to the International Classification of Headache Disorders, 3rd Edition, by a neurologist who is an expert in the field of headache will be included in the study.
Sampling Method: Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | In first enrollment, 1 minute
  The visual analog scale consists of the pain level that the person currently experiences with a vertical line on a plane. The pain felt by the person is marked as "0: no pain at all", "10: I feel very severe pain". Scoring is based on the vertical marking the participant makes for the pain he/she marks on the plane with a ruler.
Migraine Disability Assessment Questionnaire | In first enrollment, 1 minute
  Disability of migraine patients will be assessed with the Migraine Disability Assessment Questionnaire (MEDA). MEDA assesses the last 3 months of disability and consists of a 5-item self-administered test covering disability-related activities at work/school, housework, family, and social or leisure. The total number of days missed in these activities is the total score and classifies disability as minimal disability (0-5 points), mild disability (6-10 points), moderate disability (11-20 points), or severe disability (≥21).
Headache Impact Test-6 | In first enrollment, 3 minutes
  The impact of headache will be assessed with the Headache Impact Test-6 (HIT-6). HIT-6 is a quality of life questionnaire for headaches that assesses vitality, pain, psychological distress, sociability, role, and cognitive functioning. Each item is scored on a 5-point Likert scale (6=never, 8=rarely, 10=sometimes, 11=very often, 13=always). The total score is determined by summing the scores on the six items and ranges from 36 to 78 points. (≤49 = little/no impact, 50-55 = some impact, 56-59 = significant impact, and 60-78 = severe impact; higher scores indicate greater deterioration in quality of life).
Hospital Anxiety and Depression Scale | In first enrollment, 3 minutes
  Anxiety and depression will be assessed with the Hospital Anxiety and Depression Scale (HADS). 7 items of the 14-item scale assess anxiety and 7 items assess depression symptoms. It is scored between 0-3 points. By summing the subscale scores, 0-21 points can be obtained from each of the Depression and Anxiety subscales. It is stated that 0-7 points are the normal range for each subscale, 8-10 points suggest the presence of a mood disorder, and 11 and above points indicate a possible mood disorder. In addition, there are recommended cut-off scores for mild (8-10 points), moderate (11-15) and severe (16 and above) cases.

CONTACTS AND LOCATIONS:
Locations (14):
- Elite Research and Surgical Hospital, Nicosia, Cyprus
- Turkey (Türkiye) (13):
  - Bozok University, Yozgat, Merkez
  - Gazi University, Ankara, Yenimahalle
  - Mersin University, Mersin, Yenisehir
  - Ankara Atatürk Sanatoryum Training and Research Hospital, Ankara
  - Gazi University, Ankara
  - Trakya University, Edirne
  - Gaziantep City Hospital, Gaziantep
  - İstanbul University, Istanbul
  - Silivri State Hospital, Istanbul
  - Kütahya Health Sciences University, Kütahya
  - Headache and Cognition Clinic of Aynur Ozge, Mersin
  - Tokay Gaziosmanpaşa University, Tokat Province
  - Zonguldak Bülent Ecevit University, Zonguldak

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt S, Bullinger M. Current issues in cross-cultural quality of life instrument development. Arch Phys Med Rehabil. 2003 Apr;84(4 Suppl 2):S29-34. doi: 10.1053/apmr.2003.50244. PMID 12692769
- [Background] Scirepreject. The Hospital Anxiety and Depression Scale (HADS) http://www.scireproject.com/book/export/html/78.
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Aydemir Ö, Güvenir T, Küey L, Kültür S. Hastane Anksiyete ve Depresyon Ölçeğinin Türkçe formunun geçerlik ve güvenilirlik çalışması. Türk Psikiyatri Dergisi 1997;8(4):280-287
- [Background] Dikmen PY, Bozdag M, Gunes M, Kosak S, Tasdelen B, Uluduz D, Ozge A. Reliability and Validity of Turkish Version of Headache Impact Test (HIT-6) in Patients with Migraine. Noro Psikiyatr Ars. 2020 Apr 24;58(4):300-307. doi: 10.29399/npa.24956. eCollection 2021. PMID 34924791
- [Background] Kilinc HE, Oz M, Berberoglu U, Ozel Asliyuce Y, Onan D, Fanuscu A, Ulger O. Cross-cultural adaptation, reliability and validity of the Turkish version of the Henry Ford Hospital Headache Disability Inventory (HDI/T) in patients with cervicogenic headache. Disabil Rehabil. 2024 Feb;46(4):820-827. doi: 10.1080/09638288.2023.2178679. Epub 2023 Feb 14. PMID 36788454
- [Background] Ertas M, Siva A, Dalkara T, Uzuner N, Dora B, Inan L, Idiman F, Sarica Y, Selcuki D, Sirin H, Oguzhanoglu A, Irkec C, Ozmenoglu M, Ozbenli T, Ozturk M, Saip S, Neyal M, Zarifoglu M; Turkish MIDAS group. Validity and reliability of the Turkish Migraine Disability Assessment (MIDAS) questionnaire. Headache. 2004 Sep;44(8):786-93. doi: 10.1111/j.1526-4610.2004.04146.x. PMID 15330825
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Martins IP, Gouveia RG, Parreira E. Kinesiophobia in migraine. J Pain. 2006 Jun;7(6):445-51. doi: 10.1016/j.jpain.2006.01.449. PMID 16750801
- [Background] Amin FM, Aristeidou S, Baraldi C, Czapinska-Ciepiela EK, Ariadni DD, Di Lenola D, Fenech C, Kampouris K, Karagiorgis G, Braschinsky M, Linde M; European Headache Federation School of Advanced Studies (EHF-SAS). The association between migraine and physical exercise. J Headache Pain. 2018 Sep 10;19(1):83. doi: 10.1186/s10194-018-0902-y. PMID 30203180
- [Background] İdiman F. Baş ağrılarında son kırk yıl. Ş. Bıçakcı, M. Öztürk, S. Üçler, N. Karlı ve A. Siva.(Editörler). Başağrısı Tanı ve Tedavi Güncel Yaklaşımlar, Türk Nöroloji Derneği Başağrısı Çalışma Grubu Uygulamaları. 2018:9-22
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Vlaeyen JWS, Kole-Snijders AMJ, Boeren RGB, van Eek H. Fear of movement/(re)injury in chronic low back pain and its relation to behavioral performance. Pain. 1995 Sep;62(3):363-372. doi: 10.1016/0304-3959(94)00279-N. PMID 8657437
- [Background] Yilmaz, Ö. T., Yakut, Y., Uygur, F. ve Uluğ, N. (2011). Tampa Kinezyofobi Ölçeği'nin Türkçe versiyonu ve test-tekrar test güvenirliği. Fizyoterapi Rehabilitasyon, 22(1), 44-49
- [Background] Burwinkle T, Robinson JP, Turk DC. Fear of movement: factor structure of the tampa scale of kinesiophobia in patients with fibromyalgia syndrome. J Pain. 2005 Jun;6(6):384-91. doi: 10.1016/j.jpain.2005.01.355. PMID 15943960
- [Background] Kori SH, Miller RP, Todd D. Kinesophobia: a new view of chronic pain behaviour. Pain Management. 1990;3:35-43